CLINICAL TRIAL: NCT04460989
Title: Evaluation of the Impact of Customization of Total Knee Prostheses on Patient Satisfaction and Functional Outcome of Arthroplasty.
Brief Title: Assessment of Patient Satisfaction After Arthroplasty: A Comparative Study by Implant Type
Acronym: ESPACE
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00075-34; 2020-A00075-34 (Other: ANSM)
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard implant: arthroplasty with a standard implant
  Interventions: Procedure: arthroplasty
- personalized implant: arthroplasty with a customized implant
  Interventions: Procedure: arthroplasty

INTERVENTIONS:
Procedure: arthroplasty — total knee replacement

SUMMARY:
The main objective of this study is to evaluate the benefit of personalized prostheses compared to conventional prostheses on patient satisfaction 24 months after total knee arthroplasty.

DETAILED DESCRIPTION:
Prospective randomized monocentric prospective comparative study carried out as a single blind study on two parallel groups (standard implant or customized implant).

Secondary Objectives: Compare between groups :

* the functional outcome of the arthroplasty
* pain progression
* the evolution of the quality of life
* the conditions of the surgery (duration of surgery, length of hospitalization, blood loss)
* the frequency of adverse events related to arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Adult man or woman who has signed consent to participate in the study
* Patient with uni- or bilateral primary gonarthrosis
* For which an indication for total knee arthroplasty has been established

Exclusion Criteria:

* History of knee arthroplasty or osteotomy
* History of knee fracture
* Inflammatory rheumatic disease or any other progressive concomitant disease that may affect the patient's functional prognosis.
* Joint or extra-articular deformities of the lower limb of traumatic origin
* Neurological diseases, stroke sequelae
* Mental disability or any other reason that may hinder the understanding or strict application of the protocol
* Patient not affiliated to the French social security scheme
* Patient under legal protection, guardianship or trusteeship
* Patient already included in another therapeutic study protocol or having participated in another trial within the previous three months
* Arthroplasty actually performed
* Absence of per operative complications in bone (femoral or tibial bone), ligament (rupture or disinsertion of the patellar or quadricipital tendon) or nerve (lesion of the external popliteal sciatica).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with uni or bilateral primary gonarthrosis
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
IKS self-questionnaire Score at M24 | 24 MONTHS
  The score obtained on the IKS self-questionnaire at 24 months will be compared between the two treatment groups by an analysis of covariance, with the basal IKS score as a covariate and the type of prosthesis as a factor.

SECONDARY OUTCOMES:
SF12 score at M24 | 24 months
  The comparison between groups will be made on the evolution of scores, in relation to the baseline value, by an analysis of covariance with treatment and time as fixed factors, the subject as a random factor and the baseline value as a covariate. The interaction Time x Treatment will be added to the model. The effects of time and treatment will be tested at each evaluation point.
KOOS Score at M24 | 24 months
  The comparison between groups will be made on the evolution of scores, in relation to the baseline value, by an analysis of covariance with treatment and time as fixed factors, the subject as a random factor and the baseline value as a covariate. The interaction Time x Treatment will be added to the model. The effects of time and treatment will be tested at each evaluation point.
Forgotten Joint Score at M24 | 24 months
  The comparison between groups will be made on the evolution of scores, in relation to the baseline value, by an analysis of covariance with treatment and time as fixed factors, the subject as a random factor and the baseline value as a covariate. The interaction Time x Treatment will be added to the model. The effects of time and treatment will be tested at each evaluation point.

CONTACTS AND LOCATIONS:
Overall Officials: MICHEL BONNIN, MD, Principal Investigator — CENTRE ORTHOPÉDIQUE SANTY
Locations (1):
- Centre Orthopédique Santy, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beel W, Sappey-Marinier E, Latifi R; ReSurg; Ait-Si-Selmi T, Bonnin MP. Individualised compared to off-the-shelf total knee arthroplasty results in lower and less variable patellar tilt. Knee Surg Sports Traumatol Arthrosc. 2024 Dec;32(12):3163-3173. doi: 10.1002/ksa.12234. Epub 2024 Jun 12. PMID 38864165
- [Derived] Sappey-Marinier E, Beel W; ReSurg; Bonnin MP, Ait-Si-Selmi T. Better operating room efficiency and reduced staff demand: Individualised versus off-the-shelf total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2024 Dec;32(12):3174-3184. doi: 10.1002/ksa.12233. Epub 2024 Jun 12. PMID 38864156